CLINICAL TRIAL: NCT00467532
Title: A Prospective Longitudinal Study of the Effect of Burn Size on Cytomegalovirus Reactivation and Correlates of T Cell Immune Function in Patients Sustaining Significant Burn Injury
Brief Title: Effect of Burn Size on Cytomegalovirus Reactivation and Correlates of T Cell Immune Function in Burned Patients
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Bruce Cairns, MD, Medical Director, NC Jaycee Burn Center, University of North Carolina, Chapel Hill
Other Study IDs: CMV Reactivation in Burns
Record Dates: First submitted 2007-04-26; First posted 2007-04-30 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Burns; Cytomegalovirus
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the effect of burn injury on the human immune system with a focus on cytomegalovirus (CMV) reactivation and the immunologic correlates of latent viral reactivation.

Subjects will be patients admitted to the North Carolina Jaycee Burn Center with burn injury.

Blood samples will be collected over time and will be evaluated for CMV reactivation and immune cell phenotype.

DETAILED DESCRIPTION:
The purpose of this research study is to learn about infections and the immune system in people who suffer from burn injuries. The immune system changes after burn injury and infection is one of the most common complications. Cytomegalovirus (CMV) is a virus that most people are exposed to early in life; once you are exposed it lays inactive in your body forever. When the immune system is suppressed, this virus can reactivate. We would like to measure how this virus makes copies of itself in the blood stream in people with a burn injury and to look at cell markers of the immune system.

This study involves baseline and weekly blood draws for approximately 8 weeks. If blood tests show CMV infection, further monitoring of blood work may be needed after eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Burn injury,
* Positive CMV IgG level confirmative of previous CMV infection and latency.

Exclusion Criteria:

* Immunocompromising conditions including HIV/AIDS,
* End-stage renal disease,
* End-stage liver disease,
* Pregnancy,
* Rheumatologic or collagen-vascular disease requiring chronic use of steroids,
* Chronic use of immunosuppressive agents,
* Recent chemotherapy, and
* History of solid organ or allogeneic stem cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the North Carolina Jaycee Burn Center within 72 hours of burn injury with at least a 10% Total Body Surface (TBSA)burn and expected length of stay at least two weeks.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
CMV IgG and viral load PCR | Weekly until viremia resolved (negative viral load by PCR)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Cairns, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- North Carolina Jaycee Burn Center, UNC Hospitals, Chapel Hill, North Carolina, United States